CLINICAL TRIAL: NCT01468155
Title: Dabigatran for Peri Procedural Anticoagulation During Radiofrequency Ablation of Atrial Fibrillation
Brief Title: DAPPAR AF Dabigatran for Peri Procedural Anticoagulation During Radiofrequency Ablation of Atrial Fibrillation
Acronym: DAPPARAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSREB 18098
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
Keywords: PVA; peri procedural bleeding complications
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabigatran (Active Comparator): Dabigatran will be compared to historical data using other OAC methods for Pulmonary Vein Ablation
  Interventions: Drug: dabigatran

INTERVENTIONS:
Drug: dabigatran — 30 days pre ablation and 90 days post ablation
  Other Names: pradax

SUMMARY:
It is hypothesized that peri-ablation Dabigatran will be a safe and effective method of peri-procedural anticoagulation for Atrial Fibrillation (AF) ablation, resulting in a low rate of peri-procedural bleeding and thromboembolic complications.

DETAILED DESCRIPTION:
All patients will be initiated on fixed dose Dabigatran 150 mg BID at least one month prior to the ablation procedure. If patients were already on warfarin therapy, then warfarin should be stopped for a minimum of 2 days prior to Dabigatran initiation, when the INR is less than 2. Patients will remain on the same dose of Dabigatran until the day before ablation. On the day prior to ablation, patients will not take any Dabigatran, nor will any be taken on the day of ablation, until after sheath removal.

For patients in high-risk groups for bleeding, the lower dose of Dabigatran may be used, or the drug may be stopped further in advance of the procedure. For patients with age greater than 80 years old, the lower dose of Dabigatran (110 mg BID) may be used as an alternative. For patients with impaired renal function, the lower dose may be used, but the drug may be stopped earlier in advance of the procedure as per the suggestions in Appendix A.

Post-ablation, Dabigatran will be started at the same dose - either 150 mg or 110 mg - as before the ablation procedure. Dabigatran will be initiated 8 hours post sheath removal and continue twice daily until the three month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or greater.
* Patients undergoing first-time catheter ablation for AF.
* Patients with paroxysmal or persistent AF. Paroxysmal AF will be defined as self-terminating episodes less than 7 days duration. Persistent AF will be defined as episodes that last longer than 7 days duration or episodes requiring termination by electrical or chemical cardioversion.
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication. "Symptomatic" patients are those who have been aware of their AF anytime within the last 5 years prior to enrollment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of the above.
* At least one episode of AF must have been documented by ECG, Holter, loop recorder, telemetry, or transtelephonic monitoring within 24 months of entry in the trial.
* Patients must be able and willing to provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* Patients with AF felt to be secondary to an obvious reversible cause (e.g. thyroid disease, post-surgical).
* Patients with contraindications to systemic anticoagulation with heparin or a direct thrombin inhibitor.
* Patients with severe renal impairment (creatinine clearance of <30 ml/min)
* Patients with left atrial size >/= 60 mm (2D echocardiography, parasternal long axis view).
* Patients who are or may potentially be pregnant or who are not on an effective method of birth control or who are planning to get pregnant during the study.
* Patients with mechanical heart valves.
* Patients who are undergoing repeat catheter ablation of AF.
* Patients with hemorrhagic manifestations, bleeding diathesis, or patients with impairment of hemostasis.
* Lesions at risk of clinically significant bleeding - such as extensive cerebral infarction within the last 6 months, active peptic ulcer disease with recent bleeding.
* Concomitant treatment with strong P-glycoprotein inhibitors, i.e. ketoconazole.
* Known hypersensitivity to Dabigatran or Dabigatran etexilate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07-13 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
The incidence of peri-procedural major bleeding complications | 1 month prior to Pulmonary Vein Ablation and three months post ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Skanes, MD, FRCPC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Center, London, Ontario, Canada